CLINICAL TRIAL: NCT03280498
Title: Effectiveness of Ultrasonography and The Cole Formula on the Evaluation of the Appropriate Endotracheal Tube Size
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ayse Cigdem Tutuncu, MD, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 83045809
Record Dates: First submitted 2017-08-20; First posted 2017-09-12 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Intubation
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intubation with Cole formula (Other): ASA I-II pediatric patients in the age range of 2-10 years, planned to undergo elective surgeries under general anesthesia with endotracheal entubation,
  Interventions: Procedure: Intubation

INTERVENTIONS:
Procedure: Intubation — elective surgeries under general anesthesia with endotracheal entubation formula or USG asisted

SUMMARY:
In this study the effectiveness of the use of Cole formula and USG were compared in determining the number of the appropriate uncuffed ETT to be used for clinically adequate ventilation.

DETAILED DESCRIPTION:
Aim: The goal of this study was to evaluate the effectiveness of the Cole formula and ultrasonography in determining endotracheal tube size for paediatric surgery patients.

Material and methods: ASA I-II pediatric patients (n=110) in the age range of 2-10 years, planned to undergo elective surgeries under general anesthesia with endotracheal entubation, were enrolled in this study. Once patients were properly positioned after premedication and anesthesia induction, the subglottic diameter was measured using ultrasonography, and endotracheal tube (ETT) size was also calculated with the Cole formula. Subsequently patients were entubated with uncuffed ETT with sizes based on the patient's age in compliance with current clinical guide lines. To ensure adequate ventilation, the tube was replaced with an ETT of larger or smaller diameter as needed. The ETT was fastened after the placement ring had passed through the vocal cords and breath sounds were confirmed to be equal by auscultation. The size of the used ETT was compared with the size estimated from the subglottic diameter measured by ultrasonography to the size calculated with the Cole formula

ELIGIBILITY:
Inclusion Criteria:Children between 2 and 10 years of age, in the ASA I-II classification for whom elective surgery

-

Exclusion Criteria:

Children having a diagnosed syndrome, any anomaly of the upper respiratory tract and the head-neck region, recent or active upper respiratory tract infection, previous tracheastomy, requiring nasotracheal entubation, requiring surgery on an emergency basis and being in the ASA III-IV classification -

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
: The goal of this study was to evaluate the effectiveness of the Cole formula and ultrasonography in determining endotracheal tube size for paediatric surgery patients. | 12 months
  efficiency of formula

SECONDARY OUTCOMES:
To determine the correlation of weight, height and age of child with USG based endotracheal tube size, Cole formula endotracheal tube size and clinically used endotracheal tube size | 12 months
  efficiency of USG

CONTACTS AND LOCATIONS:
Locations (1):
- Cerrahpasa Medical Faculty, Istanbul, Cerrahpasa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No